CLINICAL TRIAL: NCT00464555
Title: Strategies to Improve Long Term Islet Graft Survival
Brief Title: Strategies to Improve Islet Survival
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT CIT-02
Record Dates: First submitted 2007-04-20; First posted 2007-04-23 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Allogeneic Islets; Allogeneic Islet Transplantation; Type 1 diabetes mellitus; Type 1 diabetes; T1D; T1DM; Insulin dependence; Hypoglycemia unawareness in T1D; Islet transplant; Islet transplantation; Islet graft
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Antilymphocyte Serum; Basiliximab; lisofylline; Sirolimus; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Islet Transfusion and LSF (Experimental): Participants assigned to this group will receive an islet transfusion and an immunosuppressive medication regimen containing LSF.
  Interventions: Procedure: Islet transplant; Drug: Antithymocyte globulin; Drug: Basiliximab; Drug: Lisofylline; Drug: Sirolimus; Drug: Tacrolimus

INTERVENTIONS:
Procedure: Islet transplant — Transplantation of pancreatic islet cells
Drug: Antithymocyte globulin — Immunosuppressive that selectively depletes activated T-cells and depletes resting T-cells in a dose-dependent manner.
Drug: Basiliximab — Will replace antithymocyte globulin in all islet transplantations after the first one
Drug: Lisofylline — An anti-inflammatory that may reduce the rate at which islet cells die.
Drug: Sirolimus — Maintenance immunosuppressive therapy
Drug: Tacrolimus — Maintenance immunosuppressive therapy

SUMMARY:
Type 1 diabetes is an autoimmune disease in which the insulin-producing pancreatic beta cells are destroyed, resulting in poor blood sugar control. The purpose of this study is to determine the safety and effectiveness of islet transplantation, combined with immunosuppressive medications and medications to support islet survival, for treating type 1 diabetes in individuals experiencing hypoglycemia unawareness and severe hypoglycemic episodes.

DETAILED DESCRIPTION:
Type 1 diabetes is commonly treated with the administration of insulin, either by multiple insulin injections or by a continuous supply of insulin through a wearable pump. Insulin therapy allows for long-term survival in individuals with type 1 diabetes; however, it does not guarantee constant normal blood sugar control. As a result, long-term type 1 diabetic survivors often develop vascular complications, such as diabetic retinopathy, an eye disease that can cause poor vision and blindness, and diabetic nephropathy, a kidney disease that can lead to kidney failure. Some individuals with type 1 diabetes develop hypoglycemia unawareness, a life-threatening condition that is not easily treatable with medication and is characterized by reduced or absent warning signals for hypoglycemia. For such individuals, pancreas or pancreatic islet transplantation are possible treatment options. Unfortunately, insulin independence among islet transplant recipients tends to decline over time. New strategies aimed at promoting engraftment of transplanted islets are needed to improve the clinical outcomes associated with this procedure. The purpose of this study is to determine the safety and efficacy of islet transplantation, when combined with an immunosuppressive medication regimen containing lisofylline (LSF). This regimen is intended to treat type 1 diabetes in individuals experiencing hypoglycemia unawareness and severe hypoglycemic episodes. This study will also seek to improve the understanding of determinants of success and failure of islet transplants for type 1 diabetes.

Eligible participants will be randomly assigned to this study or the Phase 3 islet transplantation study (DAIT CIT-07). Participants assigned to this study will receive LSF. Participants in this study will receive up to three separate islet transplants and a regimen of immunosuppressive medications including antithymocyte globulin (ATG) for the first transplant, sirolimus, tacrolimus, and LSF to support the engrafting of the islets into the beta-cell mass. All participants will begin receiving ATG and sirolimus 2 days prior to transplantation. ATG will be continued until 2 days post-transplant. Sirolimus will be continued for the duration of the study. All participants will also receive tacrolimus starting one day post-transplant and continuing for the duration of the study. Basiliximab will be used in place of ATG with all subsequent transplants. Participants in the LSF group will begin to receive LSF one day prior to transplant and will continue to receive LSF until 5 days post-transplant. Transplantations will involve an inpatient hospital stay and infusion of islets into a branch of the portal vein. Participants who do not achieve or maintain insulin independence by Day 75 post-transplant will be considered for a second islet transplant. Participants who remain dependent on insulin for longer than 1 month after the second transplant and who show partial graft function will be considered for a third islet transplant. Basiliximab will be used in place of ATG for the second and third transplants, if they are necessary. Participants who do not meet the criteria for a subsequent transplant and do not have a functioning graft will enter a reduced follow-up period.

There will be approximately 15 study visits following each transplant. A physical exam, review of adverse events, and blood collection will occur at most visits. A chest x-ray, abdominal ultrasound, electrocardiogram, quality of life questionnaires, urine collection, and glomerular filtration rate (GFR) testing will occur at some visits. Participants will also test their own blood glucose levels at least five times per day throughout the study. A 24-month follow-up period will take place after the participant's last transplant.

ELIGIBILITY:
Inclusion Criteria:

* Mentally stable and able to comply with study procedures
* Clinical history compatible with type 1 diabetes with onset at less than 40 years of age, insulin dependence for at least 5 years at study entry, and a sum of age and insulin dependent diabetes duration of at least 28
* Absent stimulated C-peptide (less than 0.3 ng/mL) 60 and 90 minutes post-mixed-meal tolerance test
* Involvement of intensive diabetes management, defined as:

  1. Self-monitoring of glucose values no less than a mean of three times each day averaged over each week
  2. Administration of three or more insulin injections each day or insulin pump therapy
  3. Under the direction of an endocrinologist, diabetologist, or diabetes specialist with at least three evaluations during the 12 months prior to study enrollment
* At least one episode of severe hypoglycemia in the past 12 months prior to study enrollment
* Reduced awareness of hypoglycemia. More information about this criterion, including specific definition of hypoglycemia unawareness, is in the protocol.

Exclusion Criteria:

* Body mass index (BMI) greater than 30 kg/m^2 or weight less than or equal to 50 kg
* Insulin requirement of more than 1.0 IU/kg/day or less than 15 U/day
* Hemoglobin A1C (HbA1c) greater than 10%
* Untreated proliferative diabetic retinopathy
* Systolic blood pressure higher than 160 mmHg or diastolic blood pressure higher than 100 mmHg
* Measured glomerular filtration rate (GFR) using iohexol of less than 80 mL/min/1.73m2. More information about this criterion is in the protocol.
* Presence/history of macroalbuminuria (greater than 300 mg/g creatinine)
* Presence/history of panel-reactive anti-HLA antibodies above background by flow cytometry. More information about this criterion is in the protocol.
* Pregnant, breastfeeding, or unwilling to use effective contraception throughout the study and 4 months after study completion
* Presence of history of active infection, including hepatitis B, hepatitis C, human immunodeficiency virus (HIV), or tuberculosis (TB). More information about this criterion is in the protocol.
* Negative for Epstein-Barr virus (EBV) by IgG determination
* Invasive aspergillus, histoplasmosis, or coccidioidomycosis infection within one year prior to study enrollment
* History of malignancy except for completely resected squamous or basal cell carcinoma of the skin
* Known active alcohol or substance abuse
* Baseline hemoglobin (Hgb) below the lower limits of normal, lymphopenia, neutropenia, or thrombocytopenia
* History of Factor V deficiency
* Any coagulopathy or medical condition requiring long-term anticoagulant therapy after transplantation or individuals with an INR greater than 1.5
* Severe coexisting cardiac disease, characterized by any one of the following conditions:

  1. Heart attack within the last 6 months
  2. Evidence of ischemia on functional heart exam within the year prior to study entry
  3. Left ventricular ejection fraction less than 30%
* Persistent elevation of liver function tests at the time of study entry
* Symptomatic cholecystolithiasis
* Acute or chronic pancreatitis
* Symptomatic peptic ulcer disease
* Severe unremitting diarrhea, vomiting, or other gastrointestinal disorders that could interfere with the ability to absorb oral medications
* Hyperlipidemia despite medical therapy (fasting low-density lipoprotein [LDL] cholesterol > 130 mg/dL, treated or untreated; and/or fasting triglycerides > 200 mg/dL)
* Receiving treatment for a medical condition that requires chronic use of systemic steroids, except for the use of 5 mg or less of prednisone daily, or an equivalent dose of hydrocortisone, for physiological replacement only
* Treatment with antidiabetic medication other than insulin within the past 4 weeks
* Use of any study medications within the past 4 weeks
* Received a live attenuated vaccine(s) within 2 months of enrollment
* Any medical condition that, in the opinion of the investigator, will interfere with safe participation in the trial
* Treatment with any immunosuppressive regimen at the time of enrollment
* A previous islet transplant
* A previous pancreas transplant, unless the graft failed within the first week due to thrombosis, followed by pancreatectomy and the transplant occurred more than 6 months prior to enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-12; Primary Completion 2011-11 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with insulin independence | 75 days after first transplant infusion

SECONDARY OUTCOMES:
Reduction in insulin requirements, HbA1c, mean amplitude of glycemic excursions (MAGE), glycemic lability index (LI), Ryan hypoglycemia severity (HYPO) score, fasting glucose, glucose variation, beta score | 75 days and 1 year following the first and final infusion
Quality of life measures | 75 days and 1 year following the first and final infusion, and 2 years after the final infusion

CONTACTS AND LOCATIONS:
Overall Officials: Camillo Ricordi, MD, Study Chair — Department of Surgery, University of Miami Miller School of Medicine - Diabetes Research Institute
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - University of Illinois at Chicago, Chicago, Illinois

REFERENCES:
- See also: Division of Allergy, Immunology, and Transplantation (DAIT), National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/about/organization/dait/pages/default.aspx
- See also: Click here for the Clinical Islet Transplantation Consortium Web site — http://www.citisletstudy.org